CLINICAL TRIAL: NCT05245032
Title: Biologically Focused Therapy of Treatment Refractory MDS Patients
Brief Title: Biologically Focused Therapy of Treatment-Refractory MDS Patients
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Notable Labs Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB-45236; HEMMDS0035 (Other: OnCore); IRB-45236 (Other: Stanford IRB)
Record Dates: First submitted 2022-02-09; First posted 2022-02-17 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Feasibility testing: During the screening visit, blood and/or a bone marrow sample will be obtained for the patient's standard clinical evaluation. An aliquot of the blood and/or marrow sample will be obtained for ex vivo drug sensitivity assay

SUMMARY:
This non interventional study examines the feasibility of using patient specific therapeutic screening method, ex vivo to enhance current treatment recommendations in a clinically feasible time frame of 30 days.

DETAILED DESCRIPTION:
This study utilizes the Notable Labs personalized testing service using an ex vivo assay, but does not involve actual treatment or treatment determinations. The results of these screenings will be made available to patients and their physicians for their use off study.

The primary objective of the study is:

• To determine the feasibility of selecting patient specific treatment regimens based on ex vivo within 30 days

The exploratory objectives of the study are:

• To identify biomarkers that explain ex vivo drug sensitivity results

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent;
* Myelodysplastic syndrome as defined by WHO classification (see Appendix 2), or MDS/MPN with >= 5% blasts in the bone marrow or peripheral blood, including chronic myelomonocytic leukemia (CMML) 1 and 2 by WHO classification
* Relapsed/refractory disease, defined as failed or are ineligible for hypomethylating agent therapy
* Cytogenetics reported

Exclusion Criteria:

* Hypoplastic MDS
* Patients without adequate marrow samples for ex vivo analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at a single site, namely Stanford's MDS Center.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with successful ex vivo results | 30 days
  Proportion of patients with successful ex vivo results within a 30 day period from the time marrow sample is sent to Notable Labs for ex vivo testing
Proportion of patients with successful treatment decisions | 30 days
  Proportion of patients with successful treatment decisions made by the molecular oncology board within a 30 day period from the time marrow sample is sent to Notable Labs for ex vivo testing

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Greerberg, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford MDS Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No